CLINICAL TRIAL: NCT05241730
Title: Influence of a Diet With Different Glycaemic Indices and Carbohydrate Content on Substrate Utilization, Energy Storage, and Performance-related Parameters in Endurance-trained Men
Brief Title: Glycaemic Index and Substrate Metabolism
Acronym: GI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Daniel König, Univ.-Prof. Dr. med., Head of Subunit Nutrition, Exercise and Health, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2105/2021
Record Dates: First submitted 2022-01-25; First posted 2022-02-16 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Substrate Metabolism During Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low GI (Experimental): The subjects eat 55-60 E-% carbohydrates with ≥ 65 % from low glycaemic index carbohydrates per day, the other E-% are fats and proteins.
  Interventions: Other: Training intervention; Other: Low Glycaemic Index
- High GI (Active Comparator): The subjects eat 55-60 E-% carbohydrates with ≥ 65 % from high glycaemic index carbohydrates per day, the other E-% are fats and proteins.
  Interventions: Other: Training intervention; Other: High Glycaemic Index
- Low Carb High Fat (Experimental): The subjects eat ≥ 65 E-% fats and a maximum of 50 g carbohydrates per day.
  Interventions: Other: Training intervention; Other: LCHF

INTERVENTIONS:
Other: Training intervention — The training intervention will be a 10 week training plan for endurance runners. The plan consists of five sessions per week (three basic endurance sessions and two interval sessions)
Other: High Glycaemic Index — The subjects eat 55-60 E-% carbohydrates with ≥ 65 % from high glycaemic index carbohydrates per day, the other E-% are fats and proteins.
  Arms: High GI
Other: LCHF — The subjects eat ≥ 65 E-% fats and a maximum of 50 g carbohydrates per day.
  Arms: Low Carb High Fat
Other: Low Glycaemic Index — The subjects eat 55-60 E-% carbohydrates with ≥ 65 % from low glycaemic index carbohydrates per day, the other E-% are fats and proteins.
  Arms: Low GI

SUMMARY:
Substrate metabolism during exercise can be influenced by various nutritional regimes. The effectiveness of the different nutritional regimes, which differ in their carbohydrate content, will be investigated not only by functional tests but also the measurement of the mechanistic processes in the muscle will be explored.

Magnetic resonance (MR), better known as magnetic resonance imaging (MRI), has been widely used in clinical practice as a non-invasive imaging technique. Importantly, in addition to producing anatomical images, an MR scanner also offers the possibility to measure the concentrations of a number of metabolic products. This is done through a technique known as magnetic resonance spectroscopy (MRS).

This research project asks the following questions:

* Can a diet containing carbohydrates with a low glycemic index achieve the same adaptations in basic endurance/fat metabolism as a high fat, low carbohydrate (ketogenic) diet?
* Does a high-fat, low-carbohydrate diet, compared with a high-carbohydrate diet, prevent improvements in performance in the submaximal and maximal range?
* What is the effect of diets with different carbohydrate content and variable glycemic index on endurance performance in a half marathon and a time trial?
* How do the diets with different carbohydrate content and variable glycaemic index affect the energy and glycogen stores in the muscles?

In active recreational athletes, the objectives are: (1) to investigate the effects of different diets with variable carbohydrate content and glycaemic index on substrate metabolism, (2) to determine the effects of the different diets on energy stores using multinuclear dynamic magnetic resonance spectroscopy, and (3) to measure the effects of the different diets on endurance performance.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Age between 18 and 40 years
* Recreational active in leisure time (2-3x/week physical activity)
* Motivation for performance testing and structured training plan
* Interest in different diets
* no acute or chronic illnesses

Exclusion Criteria:

* Contraindications to physical exercise according to ACSM (American College of Sports Medicine) guidelines
* Age <18 or >40 years
* Taking medication that could influence the measurements or that is prohibited in training and/or competition according to the WADA (World Anti-Doping Agency) Code
* Competitive athlete with own training plan
* Experience with intervention diets

MRI-specific exclusion criteria:

* Claustrophobia
* Cardiac pacemaker
* cochlear implant
* subcutaneous injection system
* Stents, metal implants, braces, piercings, tattoos
* Body weight of more than 180 kg or BMI of more than 37 kg/m2

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 65 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
changes in peak oxygen consumption (measured in ml/min/kg) | Baseline - 10 weeks
  VO2peak will be assessed during a graded exercise test on the treadmill.
changes in 5 km time trial (measured in mm:ss) | Baseline - 10 weeks
  5 km time trial performance will be assessed during an all out 5 km run on a 400 m running track. The time for completing the 5 km will be assessed.
changes in muscle glycogen content (measured in mmol/l muscle) | Baseline - 10 weeks
  Changes in muscle glycogen will be assessed in a thigh muscle using a MR scan.
changes in power at lactate turning point 1 (LTP1) and individual anaerobic threshold (IAS) (measured in km/h) | Baseline - 10 weeks
  Changes in power at LTP1 and IAS will be assessed during a graded exercise test on a treadmill.
changes in AUC in lactate in the graded exercise test | Baseline - 10 weeks
  Changes in AUS in lactate will be assessed during a graded exercise test on a treadmill.

SECONDARY OUTCOMES:
changes in fat free mass (measured in kg) | Baseline - 5 weeks - 10 weeks
  Changes in fat free mass will be assessed using a bioelectrical impedance analysis.
changes in fat mass (measured in kg) | Baseline - 5 weeks - 10 weeks
  Changes in fat mass will be assessed using a bioelectrical impedance analysis.
changes in skeletal muscle mass (measured in kg) | Baseline - 5 weeks - 10 weeks
  Changes in skeletal muscle mass will be assessed using a bioelectrical impedance analysis.
changes in body water (measured in l) | Baseline - 5 weeks - 10 weeks
  Changes in total and extracellular body water will be assessed using a bioelectrical impedance analysis.
changes in body weight (measured in kg) | Baseline - 5 weeks - 10 weeks
  Changes in body weight will be assessed using a bioelectrical impedance analysis.
changes in body mass index | Baseline - 5 weeks - 10 weeks
  Changes in body mass index will be assessed using a bioelectrical impedance analysis. The weight and the height will be used to calculate changes in BMI in kg/m^2.
completion time of a half marathon performance (measured in hh:mm:ss) | after 10 weeks
  The half marathon performance will be assessed during an official marathon race. The time of completion of the half marathon will be assessed.
changes in cholesterin and cholesterin subunits (measured in mg/dl) | Baseline - 10 weeks
  Changes in cholesterin and cholesterin subunits (LDL and HDL cholesterin) will be assessed with a routine blood count.
changes in rated perceived exhaustion (RPE) in 5 km time trial | Baseline - 10 weeks
  The changes in RPE will be assessed during the 5 km time trial on a running track. The RPE scale ranges from 6 to 20, where 20 means "really, really exhausting".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moitzi AM, Krssak M, Klepochova R, Triska C, Csapo R, Konig D. Effects of a 10-Week Exercise and Nutritional Intervention with Variable Dietary Carbohydrates and Glycaemic Indices on Substrate Metabolism, Glycogen Storage, and Endurance Performance in Men: A Randomized Controlled Trial. Sports Med Open. 2024 Apr 10;10(1):36. doi: 10.1186/s40798-024-00705-9. PMID 38600291